CLINICAL TRIAL: NCT07127120
Title: A Single Arm, Open Label Study to Assess the Tolerability of a Prebiotic in Adults With Parkinson's Disease and Healthy Adults
Brief Title: Open Label Single Arm Prebiotic Pilot Trial SR001
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorridi Therapeutics (Industry)
Collaborators: Illinois Institute of Technology, Chicago, USA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SR001; 1376682 (Other: WCG IRB)
Record Dates: First submitted 2025-08-08; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Parkinsons; Fiber; prebiotic; inflammation; constipation
MeSH Terms: conditions — Parkinson Disease; Inflammation; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prebiotic Fiber Bar (Experimental): Open-label consumption of prebiotic fiber bars
  1 bar/day for 4 weeks
  Interventions: Dietary Supplement: Prebiotic fiber blend

INTERVENTIONS:
Dietary Supplement: Prebiotic fiber blend — Proprietary blend of 5 prebiotic fibers and normal bar excipients Product name: NeuroFiber Dosage form: Single bar/day
  Storage conditions:
  The Study Product delivered by Sorridi to patient/subject at the beginning of study. Any remainder will be collected by Sorridi at end of study.
  Product is to be stored at room temperature in the patient's/subject's homes.
  The bar will be produced and packaged at a licensed contract manufacturer experienced in producing nutritional supplements.
  Labelling will be carried out by Sorridi Therapeutics.

SUMMARY:
The goal of this pilot clinical study is to evaluate the effect of a prebiotic fiber blend in individuals diagnosed with Parkinson's Disease. The main objectives of this pilot study are:

1. To assess the safety and tolerability of consuming 1 fiber bar/day
2. To determine if a prebiotic fiber blend impacts biological metrics and non-motor symptoms of Parkinsons Disease
3. To evaluate the effect of the fiber bar on intestinal inflammation

Participants will have blood and fecal samples collected at baseline and after 4 weeks of intervention. Participants will also complete questionnaires to monitor GI symptom severity, quality of life metrics, and Parkinson's-specific surveys. Researchers will compare biomarkers and reported assessment answers at baseline and after 4 weeks with intervention.

DETAILED DESCRIPTION:
Recent evidence has unveiled a major role of gut-brain crosstalk in the pathology of Parkinson's Disease (PD). The gastrointestinal tract is home to a diverse and complex community of microorganisms, termed the microbiota. The microbiota performs numerous functions, like digestion and metabolism of food and immune system regulation. Moreover, the microbiota produces vital molecules like neurotransmitters and metabolites that contribute to intestinal, neural, and systemic health. Dysbiosis, or an imbalanced microbiome, is common in patients with PD, and one of the major non-motor symptoms associated with PD is constipation. It is believed that an increase in pro-inflammatory bacteria and a decrease in anti-inflammatory bacteria contribute to the symptoms and pathology of PD, with recent research focusing on bacteria that produce short chain fatty acids (SCFA). SCFA are beneficial metabolites that are used as fuel by host intestinal cells, modulate inflammation, and promote overall health. Dietary fibers are the primary nutrient that is broken down by bacteria to produce SCFA. Therefore, we have formulated a prebiotic fiber blend to specifically enhance the growth and metabolism of SCFA-producing bacteria, with the aim to improve gastrointestinal health in patients with Parkinson's Disease. In this pilot clinical study, participants with PD will consume 1 fiber bar per day for 4 weeks. Questionnaires will be utilized to monitor tolerability, gastrointestinal symptoms, motor and non-motor metrics of PD. Blood and fecal samples will be collected at baseline and again after 4 weeks of consuming the fiber bar daily. The data collected during this pilot trial will be used to inform future, larger trials on the effectiveness of prebiotic fiber formulations to modulate the microbiome of PD patients, with the ultimate goal of reducing severity of PD symptoms and delaying the progression of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease by a Neurologist
* Be able to give written informed consent
* Be aged between 60-75 years
* Participants are on a stable drug regimen
* Willing to consume the study product daily for the duration of the study
* Willing to abstain from pre and probiotics for 2 weeks prior to the study and throughout the 28 days of the intervention

Exclusion Criteria:

* Participants has acute or chronic gastrointestinal disease (coeliac disease, diarrhea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers) except for hiatal hernia, gastroesophageal reflux disease, haemorrhoids.
* Participants who have consumed probiotic supplements and prebiotic supplements within 2 weeks prior to Visit 1.
* Participant suffering from severe renal disease (creatinine greater than 2.5 times normal)
* Participants with markedly abnormal liver function (alt/ast greater than 2.5 times normal)
* Plan to have a major change in dietary habits during the study.
* Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
* Participants may not be receiving treatment involving experimental drugs/supplements. If the Participant has been in a recent experimental study, these must have been completed not less than 90 days for drugs and 30 days for supplements prior to this study.
* Consumption of non-standard diet (vegetarian, vegan, gluten free, or paleo)
* Elevated bilirubin

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Tolerability of Prebiotic Fiber bar in Parkinson's Patients | From enrollment to 4 weeks on intervention
  The tolerability of consuming 1 fiber bar/day for 4 weeks. Impacts on bowel movement frequency, stool consistency (Bristol Stool Scale), gastrointestinal symptoms of bloating, cramping, flatulence will be evaluated using a GI questionnaire. Measures are reported as # of days, # of events, and severity scale of 1-4. 1=never, 2=infrequent, 3=a few times, 4=often. Values for each metric in the questionnaire will be totaled to achieve an overall GI score. A higher score is indicative of worse GI effects. A decrease in overall score will indicate improvement in GI symptoms, and will be interpreted as tolerability of prebiotic consumption.
Safety of Prebiotic Fiber bar in Parkinson's Patients | 4 weeks
  The safety of consuming 1 fiber bar/day for 4 weeks. Safety will be evaluated based on frequency of adverse events over the course of the study. Potential adverse events could include worsening of gastrointestinal distress and discomfort, changes from baseline blood metabolic measures to abnormal ranges that could indicate liver or kidney dysfunction, diabetes, etc.

SECONDARY OUTCOMES:
Changes in biomarkers of intestinal inflammation | 4 weeks
  Change in fecal calprotectin levels, as a marker of intestinal inflammation. Change in fecal zonulin levels, as a measure of gut barrier permeability.
  Both are measured in ug/g. Higher levels of calprotectin (over 50 ug/g) are indicative of gut inflammation. A decrease in the levels will be interpreted as improvement of intestinal inflammation. Higher levels of zonulin (over 110 ug/g) are indicative of more intestinal barrier permeability (leakier gut). A decrease in the levels will be interpreted as strengthening of the gut barrier.
Changes in gut microbiome composition | 4 weeks
  Changes in relative abundance and species composition of microbiome, measured in fecal samples. The microbiome will be evaluated using 16s rRNA sequencing and shotgun metagenomics.
Changes in fecal metabolites | 4 weeks
  Changes in levels of short chain fatty acids (SCFA). SCFA concentration(mmol/g) in fecal samples collected at baseline and after 4 weeks will be measured using GC/MS. Levels of individual SCFA (acetate, butyrate, propionate) as well as total levels will be compared at baseline to 4 weeks. Increases in total SCFA levels as well as increases in specific individual SCFA will be interpreted as positive impacts of the fiber formulation consumption.

OTHER OUTCOMES:
Changes in serum markers of neuroinflammation | 4 weeks
  Change in serum biomarkers of neuroinflammation: levels of neurofilament light chain (NfL) and glial fibrillary acidic protein (GFAP). Both are measured in pg/mL. High levels of NfL (over 4 pg/mL) and high levels of GFAP (over 87 pg/mL) are indicative of neurodegeneration. A decrease in levels will be interpreted as improvements in brain health and slowing of progression of neurodegeneration.
Impacts on non-motor symptoms associated with Parkinson's Disease | 4 weeks
  Changes in sleep quality, measured with the Parkinsons Disease Sleep scale (PDSS-2) questionnaire. Metrics of sleep disturbances are measured from 0-10, with 0=always and 10=never. Scores for each metric will be added together for a number total. Lower scores are indicative of more sleep disturbances, and worse symptoms. Totals will be compared from baseline to 4 weeks. Increases in total scores will be interpreted as improvements in sleep problems.
Change in symptoms of Parkinson's Disease | 4 weeks
  Changes in motor and non-motor symptoms of Parkinson's Disease will be evaluated using the MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) questionnaire. Metrics are scored from 0-4. 0=Normal or nonexistent, 1=slightly problematic, 2=mildly problematic, 3=moderately problematic, 4=severely problematic. Scores from Part I (non-motor experiences), Part II (motor experiences), Part III (motor examination), and Part IV (motor complications) will be totaled. Lower scores indicate less problematic symptoms. Totals will be compared from baseline to four weeks. Decreases in scores will be interpreted as improvements in symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sorridi Therapeutics, Northbrook, Illinois, United States

IPD SHARING:
Plan to Share IPD: No